CLINICAL TRIAL: NCT00585351
Title: Extending Acute Stroke Trials to the Aerial Inter-hospital Transfer Setting (AIRDOC)
Brief Title: Extending Acute Stroke Trials to the Aerial Inter-hospital Transfer Setting
Acronym: AIRDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: NIH 5K12RR017700-04; NIH 5K12RR017700-04
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Experimental): Advanced Notification + Ranitidine
  Interventions: Drug: Ranitidine; Other: Advanced notification
- II (Active Comparator): Advanced Notification + Placebo
  Interventions: Drug: Placebo; Other: Advanced notification
- III (Active Comparator): No advanced notification + Ranitidine
  Interventions: Drug: Ranitidine; Other: No advanced notification
- IV (Placebo Comparator): No advanced notification + Placebo
  Interventions: Drug: Placebo; Other: No advanced notification

INTERVENTIONS:
Drug: Ranitidine — 50 mg single dose injection of Ranitidine
  Arms: I; III
Drug: Placebo — 50 mg single dose injection of normal saline (placebo)
  Arms: II; IV
Other: Advanced notification — Advanced notification of study via faxed consent to local Emergency Room (ER)
  Arms: I; II
Other: No advanced notification — No advanced notification of study via faxed consent to local Emergency Room (ER)
  Arms: III; IV

SUMMARY:
We are inviting patients who have been diagnosed with an ischemic or hemorrhagic stroke and are being transferred by Air Care helicopters to the University of Iowa Hospitals and Clinics (UIHC) for further care to participate in this research study to test the following: 1) To test whether it is possible to go through all the procedures necessary to start a study, including an informed consent, before the patient is transferred by helicopter to Iowa City. 2)To test a low risk medication called, Ranitidine, that might lower the chances of developing chemical pneumonitis (irritation of the lungs by stomach contents), a fairly common complication in patients that have had a stroke. Patients will be randomly assigned to receive a single dose injection of either Ranitidine (50 milligrams (mg)) or placebo (normal saline).

DETAILED DESCRIPTION:
Ischemic or hemorrhagic stroke patients transferred by Air Care helicopters to the University of Iowa Hospitals and Clinics (UIHC) for further care will be invited to participate in a research study testing the following: 1) feasibility of beginning a research study while the patient is in transit to UIHC, and 2)test efficacy of a low risk medication called, Ranitidine, to help lower the chances of developing chemical pneumonitis in patients that have had a stroke.

Patients will be randomly assigned to receive a single dose injection of either Ranitidine (50 mg) or placebo (normal saline). Independently of the study injection, the patient will continue to receive the usual standard medical care for their stroke. The patient will be cared for by a team of doctors in the stroke service. Some of these doctors and nurses are investigators for this study and will assess the patient's neurological status to see how much the stroke has affected the patient. They will also determine by the patient's symptoms and the results of a chest x-ray (if that test becomes necessary due to fever) whether the patient has developed chemical pneumonitis They will also administer a questionnaire to the patient or their relative prior to discharge about their thoughts on doing clinical studies while being transported by the helicopter and to collect any thoughts they may have had about improving this process. Completing the questionnaire is voluntary, and the patient is free to skip any question that they would prefer to not answer.

Three months after the patient has had the stroke, they or their relative will be contacted by phone to determine the patient's long-term outcome after their stroke. After the follow-up telephone conversation the participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Presumed Ischemic stroke or intracerebral hemorrhage within past 12 hours.
* NIH Stroke Scale (NIHSS) score >/=1 point.
* Negative pregnancy test (females < 50 years old).
* No pre-stroke disability (Rankin Scale Score 0-1).
* Patient evaluated for intravenous recombinant tissue Plasminogen Activator (rtPA) and intubation by the local physicians (if appropriate).

Exclusion Criteria:

* Onset of symptoms > 12 hours or uncertain time of origin (if patient awakens with stroke, the time of onset will be the last time patient was normal).
* Reason for the transfer is to receive rtPA at the University of Iowa.
* Non-stroke etiology for symptoms.
* Temperature > 37.8 C.
* Systolic blood pressure < 100 mm Hg.
* Known allergy to ranitidine.
* White Blood Cell (WBC) > 10K.
* Hemoglobin < 9.0.
* Platelets < 100,000.
* Glucose < 60 or > 300 mg/dl.
* Current need for antibiotics.
* Terminal illness with expected survival < 3 months.
* Prison inmate or institutionalized individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique C Leira, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was from January 2007 to January 2008. Subjects recruited for this study were patients with presumed ischemic stroke or intracranial hemorrhage that were transferred to the University of Iowa Hospitals and Clinics via Air Care helicopter transport.
Groups:
- Advanced Notification: Subjects in this group are randomized to receiving advanced notification about the AIRDOC study via a telephone call and faxing of the informed consent document prior to the arrival of Air Care helicopter crew to the outside hospital where the subject is at.
- No Advanced Notification: Subjects in this group are randomized to not receiving any advanced notification about the study, so they are not provided the informed consent document until Air Care helicopter crew has arrived to the outside hospital where the subject is at.
- Advanced Notification + Consent + Not Eligible for Study Med: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of the Air Care helicopter crew to the outside hospital where the subject is at. Consent is obtained by Air Care, however, after assessments and review of records, the subject is deemed not eligible to be randomized to receive study medication.
- No Advanced Notification + Consent +Not Eligible for Study Med: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until the Air Care helicopter crew has arrived to the outside hospital where the subject is at. Consent is obtained by Air Care, however, after assessments and review of records, the subject is deemed not eligible to be randomized to receive study medication.
- Advanced Notification + Ranitidine: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of the Air Care helicopter crew to the outside hospital where the subject is at, and the subject is randomized to receiving Ranitidine.
- No Advanced Notification + Ranitidine: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until the Air Care helicopter crew has arrived to the outside hospital where the subject is at, and the subject is randomized to receiving Ranitidine.
- Advanced Notification + Placebo: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of the Air Care helicopter crew to the outside hospital where the subject is at, and the subject is randomized to receiving placebo.
- No Advanced Notification + Placebo: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until the Air Care helicopter crew has arrived to the outside hospital where the subject is at, and the subject is randomized to receiving placebo.
Period: Notification Period (Informed Consent)
Arm/Group | Advanced Notification | No Advanced Notification | Advanced Notification + Consent + Not Eligible for Study Med | No Advanced Notification + Consent +Not Eligible for Study Med | Advanced Notification + Ranitidine | No Advanced Notification + Ranitidine | Advanced Notification + Placebo | No Advanced Notification + Placebo
Started | 50 | 50 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 27 | 25 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 25 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Flight aborted | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No study medication on flight | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject refused consent for AIRDOC | 21 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Period: Enrollment Period (Intervention)
Arm/Group | Advanced Notification | No Advanced Notification | Advanced Notification + Consent + Not Eligible for Study Med | No Advanced Notification + Consent +Not Eligible for Study Med | Advanced Notification + Ranitidine | No Advanced Notification + Ranitidine | Advanced Notification + Placebo | No Advanced Notification + Placebo
Started | 0 (Please refer to additional columns for subjects in "Advanced Notification" group for this period.) | 0 (Please refer to additional columns for subjects in "No Advanced Notification" group for this period.) | 15 | 15 | 5 | 7 | 7 | 3
Completed | 0 | 0 | 15 | 15 | 3 | 5 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Unknown if alive or deceased | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Advanced Notification + Consent + Not Eligible for Study Med: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of Air Care to the outside hospital where the subject is at. Consent is obtained by Air Care, however, after assessments and review of records, the subject is deemed not eligible to be randomized to receive study medication.
- No Advanced Notification + Consent +Not Eligible for Study Med: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until Air Care has arrived to the outside hospital where the subject is at. Consent is obtained by Air Care, however, after assessments and review of records, the subject is deemed not eligible to be randomized to receive study medication.
- Advanced Notification + Ranitidine: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of Air Care to the outside hospital where the subject is at, and the subject is randomized to receiving Ranitidine.
- No Advanced Notification + Ranitidine: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until Air Care has arrived to the outside hospital where the subject is at, and the subject is randomized to receiving Ranitidine.
- Advanced Notification + Placebo: Subjects in this group are randomized to receiving advanced notification about the study via a telephone call and faxing of the informed consent document prior to the arrival of Air Care to the outside hospital where the subject is at, and the subject is randomized to receiving placebo.
- No Advanced Notification + Placebo: Subjects in this group are randomized to not receive any advanced notification about the study, so they are not provided the informed consent document until Air Care has arrived to the outside hospital where the subject is at, and the subject is randomized to receiving placebo.
- Total: Total of all reporting groups
Arm/Group | Advanced Notification + Consent + Not Eligible for Study Med | No Advanced Notification + Consent +Not Eligible for Study Med | Advanced Notification + Ranitidine | No Advanced Notification + Ranitidine | Advanced Notification + Placebo | No Advanced Notification + Placebo | Total
Number analyzed (Participants) | 15 | 15 | 5 | 7 | 7 | 3 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 2 | 4 | 4 | 1 | 25
  >=65 years | 9 | 7 | 3 | 3 | 3 | 2 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (14) | 62 (16) | 67 (13) | 62 (12) | 62 (8) | 68 (12) | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 3 | 2 | 1 | 2 | 23
  Male | 7 | 8 | 2 | 5 | 6 | 1 | 29
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 7 | 7 | 3 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Benefit of Advanced Notification in Promoting Informed Consent
Description: Number of subjects that provided informed consent for study (advanced notification vs. no advanced notification).
Time Frame: Assessed at time of enrollment into the study.
Population: Intention to treat analysis for primary outcome (number of patients consented).
Measure: Number; unit: Participants
Arm/Group | Advanced Notification | No Advanced Notification
Number analyzed (Participants) | 50 | 50
Participants | 27 | 25

2. Secondary Outcome: Prevention of Chemical Pneumonitis
Description: Number of subjects that did not develop aspiration pneumonia in the intervention group (Ranitidine vs. placebo).
Time Frame: Assessed on the day of discharge (average length of stay is approximately 3-7 days)
Population: Intention to treat analysis for secondary outcome (number of participants with aspiration pneumonia).
Measure: Number; unit: Participants
Arm/Group | Advanced Notification + Ranitidine | No Advanced Notification + Ranitidine | Advanced Notification + Placebo | No Advanced Notification + Placebo
Number analyzed (Participants) | 5 | 7 | 7 | 3
Participants | 5 | 7 | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were reported to the investigator within 24 hours of acknowledgment. Serious Adverse Events were reported to the IRB within 24-72 hours.
Description: AE not collected for X groups.
Arm/Group | Advanced Notification + Consent + Not Eligible for Study Med | No Advanced Notification + Consent +Not Eligible for Study Med | Advanced Notification + Ranitidine | No Advanced Notification + Ranitidine | Advanced Notification + Placebo | No Advanced Notification + Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/5 | 0/7 | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/5 | 0/7 | 1/7 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Notification + Consent + Not Eligible for Study Med (N=15) | No Advanced Notification + Consent +Not Eligible for Study Med (N=15) | Advanced Notification + Ranitidine (N=5) | No Advanced Notification + Ranitidine (N=7) | Advanced Notification + Placebo (N=7) | No Advanced Notification + Placebo (N=3)
Subarachnoid Hemorrhage (SAH) resulting in Death (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject was randomized to Advanced Notification + Ranitidine. Subject's admitting diagnosis was SAH. Did receive study drug, but did not improve, so family pursued palliative care and subject passed away. Event deemed not related to study drug.
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject was randomized to Advanced Notification + Placebo. Subject's admitting diagnosis was intracranial hemorrhage, and had myocardial infarction. Received study drug, but passed away from cardiac arrest. Event deemed not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Notification + Consent + Not Eligible for Study Med (N=15) | No Advanced Notification + Consent +Not Eligible for Study Med (N=15) | Advanced Notification + Ranitidine (N=5) | No Advanced Notification + Ranitidine (N=7) | Advanced Notification + Placebo (N=7) | No Advanced Notification + Placebo (N=3)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One subject in the advanced notification + placebo group developed aspiration pneumonia.

LIMITATIONS AND CAVEATS:
Some procedural errors by the helicopter crew at the start of the trial, reliability of the stroke diagnosis from the outside hospital, and the possibility for a lower consent rate if a higher risk profile medication were used instead of Ranitidine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No